CLINICAL TRIAL: NCT00189605
Title: Prospective, Randomized, Multi-center Clinical Study of Plasma Disc Decompression Efficacy
Brief Title: Prospective, Randomized, Multi-center Clinical Study of Plasma Disc Decompression
Acronym: SPINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ArthroCare Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-704LB
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Radicular Pain
Keywords: Plasma disc decompression; Intradiscal Pressure; Steroid Injection; Epidural Steroid Injection; Selective Nerve Root Injection; Leg Pain; Radicular Pain; Coblation; SNRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Fluoroscopy guided transforaminal epidural steroid injection (TFESI)
  Interventions: Drug: Fluoroscopy guided transforaminal epidural steroid injection (TFESI)
- 2 (Experimental): Percutaneous Disc Decompression of the lumbar level which is secondary to radicular pain
  Interventions: Device: Perc-DLR/Perc-DLG

INTERVENTIONS:
Device: Perc-DLR/Perc-DLG — Device technique will be used per IFU
  Other Names: Percutaneous Disc Decompression
  Arms: 2
Drug: Fluoroscopy guided transforaminal epidural steroid injection (TFESI) — Injection of steroid solution into the lumbar level
  Other Names: TFESI
  Arms: 1

SUMMARY:
The goal of this post-marketing surveillance study is to compare two procedures which are used to treat patients who require a disc decompression procedure. These procedures are: 1) plasma disc decompression procedure using Coblation technology and 2) fluoroscopy guided transforaminal epidural steroid injection (TFESI). The study will evaluate treatment efficacy and rate of improvement in symptoms through the first six months following the procedure.

The principal objectives of this study are to determine whether subjects receiving the plasma disc decompression procedure demonstrate:

1. Improved clinical outcomes over subjects receiving TFESI
2. More rapid reversal of symptoms than subjects receiving TFESI

DETAILED DESCRIPTION:
Chronic leg and back pain are two of the most common ailments in our society, and are associated with serious financial and social consequences. One surgical treatment modality is plasma disc decompression, based on the principle that inducing a small reduction of volume in the closed hydraulic space of an intact (contained herniated) disc can relieve pressure, and thereby reduce or eliminate pain. Another widely accepted treatment is transforaminal epidural steroid injection (TFESI), which delivers a high concentration of corticosteroid to the targeted disc nerve interface, and is thought to decrease pain by reducing inflammation.

This study proposes to compare the efficacy of the plasma disc decompression procedure to the standard TFESI series in patients who have failed to improve after an initial TFESI injection. The goal is to better understand the differences between these two treatment modalities and to monitor the rates of symptom improvement through the first six months between patients receiving a series of at least two selective nerve root injections and those undergoing the one-time plasma disc decompression procedure after failing one fluoroscopy guided TFESI. Patients will continue to be monitored over the 2-year post-procedure period to assess stability of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has one symptomatic contained, focal herniated lumbar disc.
2. Patient's age should be at least 18 years old and no more than 75 years old.
3. Selective nerve root injection or epidural steroid injection for symptomatic herniated disc, received between 3 weeks and six months ago.
4. A VAS score for radicular pain of 50 or greater on a scale of 0 to 100.
5. Radicular pain concordant with image findings (MRI or CT).
6. Disc height greater than 50%.
7. Patient signs informed consent.

Exclusion Criteria:

1. Patient is pregnant, or pregnancy is suspected or planned within the study timeframe.
2. Patient is receiving Worker's compensation or is in litigation related to back/leg pain.
3. Patient has a cardiac pacemaker, automatic defibrillator, or any peripheral stimulator leads in the lumbar area.
4. Allergy to contrast media or drugs to be used in the intended procedure.
5. Medical co-morbidities that preclude surgical intervention.
6. Patient is receiving anti-psychotic therapy.
7. Patient is a prisoner.
8. Patient is incapable of understanding or responding to the study questionnaires.
9. History of previous spinal surgery at, or directly adjacent to, the level to be treated.
10. Patient is morbidly obese (BMI ≥ 40).
11. Patient is simultaneously participating in another device or drug study related to limb/axial pain.
12. Patient has a spinal fracture, tumor or infection.
13. Radicular pain originating from more than one disc level.
14. Axial (back) pain greater than radicular (leg) pain.
15. Clinical evidence of cauda equina syndrome.
16. Progressive neurologic deficit.
17. Radiological evidence of spondylolisthesis at the level to be treated.
18. Radiological evidence of moderate/severe stenosis at the level to be treated.
19. Evidence of extruded or sequestered disc herniation on magnetic resonance imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pain status change assessed using a visual analogue scale (VAS) for radicular pain intensity. | 6 weeks, 3 mos., 6 mos., 1 year, 2 years

SECONDARY OUTCOMES:
Functional status change evaluated using the Oswestry Disability Questionnaire. | 6 weeks, 3 mos., 6 mos., 1 year, 2 years
General health status change determined using the SF-36. | 6 weeks, 3 mos., 6 mos., 1 year, 2 years
Employment status change examined using a questionnaire developed by the American Academy of Orthopaedic Surgeons (AAOS) and the North American Spine Society (NASS). | 6 weeks, 3 mos., 6 mos., 1 year, 2 years
Subject global satisfaction post-procedure assessed using a global satisfaction statement. | 6 weeks, 3 mos., 6 mos., 1 year, 2 years
Change in frequency and type of pain medication use. | 6 weeks, 3 mos., 6 mos., 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gerzten, MD, Principal Investigator — Univ. of Pittsburgh Medical Center
Locations (13):
- United States (13):
  - The Orthopedic Clinic Association, Scottsdale, Arizona
  - Innovative Spine Care, Little Rock, Arkansas
  - SpectrumCare Rehabilitation Medical Center Inc., Napa, California
  - North Valley Rehabilitation Hospital, Thornton, Colorado
  - Beth Israel Deaconess Medical Center, Arnold Pain Management Center,, Boston, Massachusetts
  - The University of Michigan, The Spine Program, Ann Arbor, Michigan
  - Medical Advanced Pain Specialists (MAPS), Edina, Minnesota
  - TRIA Orthropaedic Center, Minneapolis, Minnesota
  - OrthoCarolina, Charlotte, North Carolina
  - University of Pittsburgh Medical Center (UPMC) Presbyterian, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Consultants in Pain Research, San Antonio, Texas
  - University of Vermont College of Medicine, Center for Pain Mgmt, Burlington, Vermont